CLINICAL TRIAL: NCT04617678
Title: A Comprehensive Approach to Head and Neck Cancer Prehabilitation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sanford Health (Other)
Collaborators: University of North Dakota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CTR H&N Cancer Prehab
Record Dates: First submitted 2020-10-23; First posted 2020-11-05 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cancer of Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Non-randomized prospective two-arm clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Prospective Prehabilitation (Active Comparator): Prospectively enrolling patients into a prehabilitation program for head and neck cancer.
  Interventions: Other: Prehabilitation Program
- Prospective Control (No Intervention): Prospectively enrolling patients to a control arm with no intervention.

INTERVENTIONS:
Other: Prehabilitation Program — We will assess whether prehabilitation intervention helps mitigate adverse symptoms (e.g., anxiety, depression, suicidality, distress, nutritional status, dysphagia, sarcopenia, and well-being) on a sample of head and neck cancer patients. Subjects will attend a Prepare for Surgery Heal Faster session and meet with a physical therapist, registered dietician, speech language pathologist, and masters of social work at pre-treatment, 6-8 weeks post-treatment, and 5-6 months post-treatment completion.
  Arms: Prospective Prehabilitation

SUMMARY:
Head and neck cancer accounts for 3% of malignancies in the United States. However, the diagnosis and treatment for head and neck cancer is considered to be debilitating. Not because of its morbidity, but due to the extremely rigorous treatment course which has a profound impact on patients physical, social, and emotional functioning. Disfigurement and sensorimotor deficits further compound this impact. Head and neck cancer patients contend with treatments that can significantly affect their quality of life. Treatment regularly results in decreased functional capacity and decreased quality of life. Physical impairments are manifested through, but not limited to, disfigurement, deconditioning, communication issues, "swallowing, speech, breathing, and cancer-related fatigue". Premorbid factors such as preexisting anxiety and depression, chemical dependency, financial barriers, and lack of social support system are unique obstacles to the head and neck cancer population impacting treatment and outcomes. Due to these factors, patients experience higher rates of anxiety and depression, psychological distress, and fear of cancer recurrence. In fact, "compared with other survivors of cancer, head and neck cancer survivors are almost 2 times more likely to die from suicide". In view of the aforementioned research, Roger Maris Cancer Center's head and neck cancer will implement a prehabilitation program that evaluates each patient using standardized screening tools and provide personalized education and interventions. This project evaluates a more comprehensive and proactive multidisciplinary approach to improve treatment and outcomes in head and neck cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Equal to or greater than 18 years of age
* Diagnosis of head and neck cancer
* Actively pursuing cancer treatment with a curative intent
* Willing and able to provide written consent

Exclusion Criteria:

* Patients with cardiac arrhythmia with implanted pacemaker
* Patients with other implanted electronic equipment/device
* Patients undergoing external defibrillation
* Pregnant women (per BIS instructions for use, pregnant women should not participate)
* Patient weight exceeding 375 lbs.
* Patient has a metal allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10-21 (Actual); Primary Completion 2025-12-05 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Difference between treatment and control group, from baseline in the BHS-6 to after treatment. | Baseline; post-treatment, ranging from 2 weeks to 6 months; and 6-months follow-up
  The Behavioral Health Screening 6 (BHS-6) is a validated, self-report instrument assessing psychological health. Higher scores indicate greater psychological distress. Difference = (Treatment score - Control score).
Difference between treatment and control group, from baseline in the C-SSRS to after treatment. | Baseline; post-treatment, ranging from 2 weeks to 6 months; and 6-months follow-up
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is a validated, self-report instrument assessing suicidality. Higher scores indicate greater suicidality. Difference = (Treatment score - Control score).
Difference between treatment and control group, from baseline in the NCCN Distress Thermometer after treatment. | Baseline; post-treatment, ranging from 2 weeks to 6 months; and 6-months follow-up
  The National Comprehensive Cancer Network (NCCN) Distress Thermometer is a validated, self-report instrument assessing psychological health. Higher scores indicate greater psychological distress. Difference = (Treatment score - Control score).
Difference between treatment and control group, from baseline in the MDADI to after treatment. | Baseline; post-treatment, ranging from 2 weeks to 6 months; and 6-months follow-up
  The MD Anderson Dysphagia Inventory (MDADI) is a validated, self-report instrument of functional assessments of dysphasia and overall functioning. Higher scores indicate better quality of life and higher day-to-day functioning. Difference = (Treatment score - Control score).
Difference between treatment and control group, from baseline in the FACT-H&N (Version 4) to after treatment. | Baseline; post-treatment, ranging from 2 weeks to 6 months; and 6-months follow-up
  The FACT-H&N (Version 4) is a validated, self-report instrument of functional assessments of dysphasia and overall functioning. Higher scores indicate better quality of life and higher day-to-day functioning. Difference = (Treatment score - Control score).

SECONDARY OUTCOMES:
Impact of sarcopenia on functioning | Baseline; post-treatment, ranging from 2 weeks to 6 months
  Sarcopenia will be measured using bioimpedence spectroscopy technology (BIS), a validated noninvasive measure of volume of fluids in various parts of the body. Functional assessments (sit to stand, grip strength, and two-minute walk test) will be tested as possible predictors of sarcopenia.
Difference between treatment and control group on sarcopenia measures | Post-treatment, ranging from 2 weeks to 6 months
  Sarcopenia measures collected via computed tomography will be used to compare patients who completed the prehabilitation program and those who have not.
Change from baseline to after treatment on the BHS-6. | Baseline; post-treatment, ranging from 2 weeks to 6 months; 6 months follow-up
  The Behavioral Health Screening 6 (BHS-6) is a validated self-report measure of psychological health, with higher scores indicating greater psychological distress. Change = (Post-treatment score - Baseline score).
Change from baseline to after treatment on the C-SSRS. | Baseline; post-treatment, ranging from 2 weeks to 6 months; 6 months follow-up
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is a validated self-report measure of psychological health, with higher scores indicating greater psychological distress. Change = (Post-treatment score - Baseline score).
Change from baseline to after treatment on the NCCN Distress Thermometer. | Baseline; post-treatment, ranging from 2 weeks to 6 months; 6 months follow-up
  The National Comprehensive Cancer Network (NCCN) Distress Thermometer is a validated self-report measure of psychological health, with higher scores indicating greater psychological distress. Change = (Post-treatment score - Baseline score).
Change from baseline to after treatment on the 2-min walk test. | Baseline; post-treatment, ranging from 2 weeks to 6 months; 6 months follow-up
  The 2-min walk test is a validated objective measure of physical functioning. Change = (Post-treatment score - Baseline score).
Change from baseline to after treatment on the 30 seconds sit to stand. | Baseline; post-treatment, ranging from 2 weeks to 6 months; 6 months follow-up
  The 30 seconds sit to stand is a validated objective measure of physical functioning. Change = (Post-treatment score - Baseline score).
Change from baseline to after treatment on the grip strength. | Baseline; post-treatment, ranging from 2 weeks to 6 months; 6 months follow-up
  The grip strength is a validated objective measure of physical functioning. Change = (Post-treatment score - Baseline score).
Change from baseline to after treatment on the NFPE. | Baseline; post-treatment, ranging from 2 weeks to 6 months; 6 months follow-up
  The Nutrition Focused Physical Exam (NFPE) is a validated objective measure of physical functioning. Change = (Post-treatment score - Baseline score).
Change from baseline to after treatment on the MDADI. | Baseline; post-treatment, ranging from 2 weeks to 6 months; 6 months follow-up
  The MD Anderson Dysphagia Inventory (MDADI) is a validated, self-report instrument of functional assessments of dysphasia and overall functioning. Higher scores indicate better quality of life and higher day-to-day functioning. Change = (Post-treatment score - Baseline score).
Change from baseline to after treatment on the BIS. | Baseline; post-treatment, ranging from 2 weeks to 6 months; 6 months follow-up
  The Bioelectic impedance spectroscopy (BIS) is a validated objective measure of physical functioning. Change = (Post-treatment score - Baseline score).
Change from baseline to after treatment on the FACT-H&N (Version 4). | Baseline; post-treatment, ranging from 2 weeks to 6 months; 6 months follow-up
  The FACT-H&N (Version 4) is a validated, self-report instrument of functional assessments of overall functioning. Higher scores indicate better quality of life and higher day-to-day functioning. Change = (Post-treatment score - Baseline score).

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Hysjulien, PsyD, Principal Investigator — Sanford Health
Locations (2):
- United States (2):
  - Sanford Health, Fargo, North Dakota
  - Sanford Health, Sioux Falls, South Dakota

REFERENCES:
- [Background] Samuel SR, Maiya AG, Fernandes DJ, Guddattu V, Saxena PUP, Kurian JR, Lin PJ, Mustian KM. Effectiveness of exercise-based rehabilitation on functional capacity and quality of life in head and neck cancer patients receiving chemo-radiotherapy. Support Care Cancer. 2019 Oct;27(10):3913-3920. doi: 10.1007/s00520-019-04750-z. Epub 2019 Mar 27. PMID 30919154
- [Background] Stenson, K. M. (2019). Epidemiology and risk factors for head and neck cancer. UpToDate. Retrieved, November 15, 2019 from https://www.uptodate.com/contents/epidemiology-and-risk-factors-for-head-and-neck-cancer.
- [Background] Osazuwa-Peters N, Simpson MC, Zhao L, Boakye EA, Olomukoro SI, Deshields T, Loux TM, Varvares MA, Schootman M. Suicide risk among cancer survivors: Head and neck versus other cancers. Cancer. 2018 Oct 15;124(20):4072-4079. doi: 10.1002/cncr.31675. Epub 2018 Oct 18. PMID 30335190
- [Background] Beck ACC, Passchier E, Retel VP, Stuiver MM, van der Molen L, Klop WMC, Navran A, van Harten WH, van den Brekel MWM. Study protocol of a prospective multicenter study comparing (cost-)effectiveness of a tailored interdisciplinary head and neck rehabilitation program to usual supportive care for patients treated with concomitant chemo- or bioradiotherapy. BMC Cancer. 2019 Jul 3;19(1):655. doi: 10.1186/s12885-019-5874-z. PMID 31269918
- [Background] Jung AR, Roh JL, Kim JS, Kim SB, Choi SH, Nam SY, Kim SY. Prognostic value of body composition on recurrence and survival of advanced-stage head and neck cancer. Eur J Cancer. 2019 Jul;116:98-106. doi: 10.1016/j.ejca.2019.05.006. Epub 2019 Jun 10. PMID 31185387
- [Background] Barrett-Bernstein M, Carli F, Gamsa A, Scheede-Bergdahl C, Minnella E, Ramanakumar AV, Tourian L. Depression and functional status in colorectal cancer patients awaiting surgery: Impact of a multimodal prehabilitation program. Health Psychol. 2019 Oct;38(10):900-909. doi: 10.1037/hea0000781. Epub 2019 Aug 5. PMID 31380686
- [Background] Chen AY, Frankowski R, Bishop-Leone J, Hebert T, Leyk S, Lewin J, Goepfert H. The development and validation of a dysphagia-specific quality-of-life questionnaire for patients with head and neck cancer: the M. D. Anderson dysphagia inventory. Arch Otolaryngol Head Neck Surg. 2001 Jul;127(7):870-6. PMID 11448365
- [Background] D'Antonio LL, Zimmerman GJ, Cella DF, Long SA. Quality of life and functional status measures in patients with head and neck cancer. Arch Otolaryngol Head Neck Surg. 1996 May;122(5):482-7. doi: 10.1001/archotol.1996.01890170018005. PMID 8615964
- [Background] List MA, D'Antonio LL, Cella DF, Siston A, Mumby P, Haraf D, Vokes E. The Performance Status Scale for Head and Neck Cancer Patients and the Functional Assessment of Cancer Therapy-Head and Neck Scale. A study of utility and validity. Cancer. 1996 Jun 1;77(11):2294-301. doi: 10.1002/(SICI)1097-0142(19960601)77:113.0.CO;2-S. PMID 8635098
- [Background] Minnella EM, Awasthi R, Loiselle SE, Agnihotram RV, Ferri LE, Carli F. Effect of Exercise and Nutrition Prehabilitation on Functional Capacity in Esophagogastric Cancer Surgery: A Randomized Clinical Trial. JAMA Surg. 2018 Dec 1;153(12):1081-1089. doi: 10.1001/jamasurg.2018.1645. PMID 30193337
- [Background] Mordarski BA, Hand RK, Wolff J, Steiber AL. Increased Knowledge, Self-Reported Comfort, and Malnutrition Diagnosis and Reimbursement as a Result of the Nutrition-Focused Physical Exam Hands-On Training Workshop. J Acad Nutr Diet. 2017 Nov;117(11):1822-1828. doi: 10.1016/j.jand.2017.06.362. Epub 2017 Aug 16. No abstract available. PMID 28821385
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Sealy MJ, Dechaphunkul T, van der Schans CP, Krijnen WP, Roodenburg JLN, Walker J, Jager-Wittenaar H, Baracos VE. Low muscle mass is associated with early termination of chemotherapy related to toxicity in patients with head and neck cancer. Clin Nutr. 2020 Feb;39(2):501-509. doi: 10.1016/j.clnu.2019.02.029. Epub 2019 Feb 22. PMID 30846324
- [Background] Wall LR, Ward EC, Cartmill B, Hill AJ. Physiological changes to the swallowing mechanism following (chemo)radiotherapy for head and neck cancer: a systematic review. Dysphagia. 2013 Dec;28(4):481-493. doi: 10.1007/s00455-013-9491-8. PMID 24078216